CLINICAL TRIAL: NCT02483494
Title: Effectiveness of Advanced Practice Nurse-Led Telehealth on Readmissions and Health Related Outcomes Amongst Patients Post Acute Myocardial Infarction: ALTRA Study
Brief Title: Effectiveness of Advanced Practice Nurse-Led Telehealth on Readmissions
Acronym: ALTRA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Heart Centre, Singapore (Other)
Collaborators: National University Hospital, Singapore (Other)
Responsible Party: Principal Investigator, Karen Koh, Assistant Director of Nursing, National University Heart Centre, Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2014\00793; RG2013/03 (Other Grant/Funding Number: Singapore Heart Foundation)
Record Dates: First submitted 2015-06-23; First posted 2015-06-29 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Acute Myocardial Infarction; Acute Coronary Syndrome
Keywords: Telemedicine; Advanced Practice Nurse
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- APN-led Telemedicine (Experimental): Participants will receive APN-led Telemedicine in addition to usual care.
  Interventions: Other: APN-led Telemedicine
- Usual care (No Intervention): Participants will receive the standard of care which includes education by cardiac care nurses and face-to-face consultations.

INTERVENTIONS:
Other: APN-led Telemedicine — Allocation to experimental or Usual care is 1:1.
  The four study APNs will be delivering the care and have at least three years working experiences in coronary care settings. A telephonic script and study protocol is made available to ensure standardization of intervention.
  Arms: APN-led Telemedicine

SUMMARY:
Aim. To develop and examine the effectiveness of an APN-led telehealth rehabilitative programme as a transitional nursing therapeutic on readmission rates and health related outcomes amongst patients with Acute Myocardial Infarction (AMI) post discharge.

Design. Randomized controlled trial with repeated measures.

Methodology. A consecutive sampling of 172 patients with AMI will be recruited from a tertiary hospital in Singapore. Participants will be randomised into two groups. The experimental group (ALTRA) will receive APN-led telehealth rehabilitative programme upon discharge in addition to standard care. The control group will receive only standard follow-up care.

DETAILED DESCRIPTION:
Ischaemic heart disease is the third leading cause both for death and illness for hospitalisation in Singapore. Epidemiological data shows that the incidence of acute myocardial infarction (AMI) stands around 7000 plus in Singapore. In United States, nearly 20% of patients with AMI are readmitted within 30 days of discharge causing the healthcare system a huge financial burden. These readmissions have been shown to be associated with lower patient satisfaction and less inefficient healthcare.

Cardiac rehabilitation has been proven to be an effective strategy in improving quality of life and reducing readmission. However, this structured programme which comprise of clinical review, education and exercise, has poor uptake rate for varied reasons. It is important that newer strategies are being explored and developed to cater to the changing needs of the patient population. One of which is to utilize telemedicine with combination of Advanced Practice Nurse delivering the care remotely.

This is a substudy of IMMACULATE STUDY (NCT02468349) where more details can be found.

ELIGIBILITY:
Inclusion Criteria:

* Typical history of ischemic chest pain or angina equivalent symptoms (e.g. acute onset dyspnea)> 30 minutes
* Undergone PCI for index event
* NT-Pro-BNP ≥1000 ng/L
* Cinically diagnosed AMI at high risk of ventricular remodeling (STEMI or NSTEMI):

(Anterior or large inferior STEMI)

* ECG changes>0.1mV ST segment elevation in two or more contiguous limb leads or precordial leads or
* Presence of pathological Q waves in two or more contiguous limb leads or precordial leads.
* Typical rise or fall of cardiac enzymes (cardiac troponin value exceeding the 99th percentile).
* Angiographic findings of proximal/mid LAD, proximal LCX or RCA occlusion for STEMI.

(Or NSTEMI with)

* Typical rise or fall of cardiac enzymes (cTn value exceeding the 99th percentile).
* Peak cTnI should be >10ug/L, TnT-hs>250 ng/L or CK-MB >80 IU/L
* LVEF (echocardiography) ≤ 40% or Kilip class ≥2

Exclusion Criteria:

* Hypersensitivity to ticagrelor, aspirin or any excipients
* Active pathological bleeding
* History of intracranial haemorrhage
* Infection within 6 weeks preceding the primary angioplasty, inflammatory disorders, Hepatitis, HIV, autoimmune disease or on immunosuppressive therapy
* Women of childbearing potential, known to be pregnant, breast-feeding, or intend to become pregnant during the study period.
* History of non-ischaemic cardiomyopathy or malignancy
* History of significant valvular heart disease (moderate or severe MS, MR, AS, AR, TR)
* Planned CABG within the next 6 weeks
* Cardiogenic shock unable to be weaned off inotropes or IABP
* Asthma or any other contraindications to beta-blockers
* Arrhythmias precluding proper CMR image acquisition, including atrial fibrillation and frequent atrial or ventricular ectopy of > 1 in 5 intrinsic ECG complexes
* Contraindications to cardiac magnetic resonance imaging including claustrophobia, pacemaker or ICD implantation, mechanical valve or other metallic implants
* Significant liver impairment
* Renal impairment (eGFR<45 ml min -1), end stage renal failure on renal replacement therapy
* Anaemia (Hb<10 g/dL)
* Psychosocial barriers to telemedicine adoption (screening for education level, dementia, substance abuse and other psychological disorders)
* Participants who cannot be followed up
* Participants not able or willing to consent for study

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2015-07-08 (Actual); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
Readmissions Days | 30 days
  Cardiac and non-cardiac causes Readmission days per 1000 follow up days will be calculated using the total number of sample in that arm x follow days (i.e. 30 days in this instance) as the denominator. (Please refer to references attached)

SECONDARY OUTCOMES:
Readmissions Days Per 1000 follow up days | 6 months
  Cardiac and non-cardiac causes
ED visits or unplanned self-reported doctor visits | 6 months
  Cardiac and non-cardiac causes
Cardiac Self-Efficacy Scale | 6 months
  Health Related Outcomes
Myocardial Infarction Dimension Assessment Scale | 6 months
  Health Related Outcomes
EuroQoL | 6 months
  Health Related Outcomes
Hospital Anxiety and Depression Scale | 6 months
  Health Related Outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Karen Koh, Principal Investigator — National University Heart Centre, Singapore; A Mark Richards, Study Chair — National University Heart Centre, Singapore; Mark Chan, Principal Investigator — National University Heart Centre, Singapore
Locations (1):
- National University Hospital, Kent Ridge, Singapore

REFERENCES:
- [Background] Young W, Rewa G, Goodman SG, Jaglal SB, Cash L, Lefkowitz C, Coyte PC. Evaluation of a community-based inner-city disease management program for postmyocardial infarction patients: a randomized controlled trial. CMAJ. 2003 Oct 28;169(9):905-10. PMID 14581307
- [Derived] Koh KW, Wang W, Richards AM, Chan MY, Cheng KK. Effectiveness of advanced practice nurse-led telehealth on readmissions and health-related outcomes among patients with post-acute myocardial infarction: ALTRA Study Protocol. J Adv Nurs. 2016 Jun;72(6):1357-67. doi: 10.1111/jan.12933. Epub 2016 Feb 25. PMID 26915719